CLINICAL TRIAL: NCT00570947
Title: CPR Prescription Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh Valley Hospital (Other)
Responsible Party: Principal Investigator, Marna Rayl Greenberg, Director of Emergency Medicine Research, Lehigh Valley Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2-20070910
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Prevention of Sudden Death
Keywords: CPR Anytime

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Class (Active Comparator): The control group will be advised to take a traditional CPR class and be offered a list of local classes.
  Interventions: Other: CPR Anytime Kit

INTERVENTIONS:
Other: CPR Anytime Kit — The study group will be asked to fill the CPR Anytime ™ prescription and complete the program. They will be encouraged to include other friends and family members in the program

SUMMARY:
In this study we hope to show that prescriptions provided for CPR Anytime™ to patients who are at risk for or have heart disease at three key locations, can motivate families to learn the skill. We will use our ED sites, an office based primary care setting, and an office based cardiology practice. Participants will be given the pharmacy locations where they can be purchased. Optimally they will complete the program at home with their family.

Research Hypothesis:

1. Families of patients at risk for coronary artery disease can be motivated to learn CPR by receiving a prescription for a CPR Anytime ™ self learning kit.
2. As part of the multiplier effect, an additional 1.5 family members per participant are projected to be trained to perform CPR.
3. Families may experience a "teachable moment" when their loved one is in the emergency department. In comparison to the office settings, this may increase the likelihood that they fill the prescription for CPR Anytime® and complete the learning kit.

DETAILED DESCRIPTION:
This will be a prospective study of patients presenting to one of three recruiting sites (emergency department and office based primary care/cardiology settings). Physicians at all settings will agree to be a part of the Physician CPR Prescription program. Participating physicians are provided with a description of the Physician CPR Prescription program and pre-printed CPR prescription pads. The front side of the prescription is preprinted with the information needed to obtain CPR Anytime ™ for Friends and Family. The back of the prescription is preprinted with "Quick Facts" to assist the physician in delivering a consistent and persuasive CPR message to patients and their families.

After consent, participants will be randomized to one of two groups. The control group will be advised to take a traditional CPR class and be offered a list of local classes. Phone follow up at approximately 3 months will assess their participation. The study group will be asked to fill the CPR Anytime ™ prescription and complete the program. They will be encouraged to include other friends and family members in the program. Follow up phone survey at approximately three months will assess compliance with physician recommendations to fill the prescription, as well as actual completion of the materials (and possible multiplier effect).

Comparisons between the sites regarding efficacy of prescribing will be performed. Results will be reported as mean +/- standard deviation, % or frequencies to summarize patient characteristics. One way ANOVA will be used to compare the three groups for continuous data and chi-square for categorical data.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* 45 or older
* Competent outpatient.
* Have DVD access in home.
* Willing to fill prescriptions at Spectrum pharmacy.
* Never had CPR, or CPR greater than 1 year ago.
* Have a risk factor for heart disease or have heart disease.

Exclusion Criteria:

* Non English speaking
* Minors
* Incompetent or significantly ill/distressed
* No DVD access
* Unwilling to fill rx at spectrum.
* CPR less than 1 year ago.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2007-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Completion of CPR | 3 months

SECONDARY OUTCOMES:
Family Member completion of CPR | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marna R Greenberg, D.O., Principal Investigator — LVH